CLINICAL TRIAL: NCT02716818
Title: A Phase III Study of Efficacy, Safety and Tolerability of Chronocort® Compared With Standard Glucocorticoid Replacement Therapy in the Treatment of Congenital Adrenal Hyperplasia
Brief Title: Comparison of Chronocort® With Standard Glucocorticoid Therapy in Patients With Congenital Adrenal Hyperplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIUR-005
Record Dates: First submitted 2016-02-26; First posted 2016-03-23 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: Glucocorticoid therapy
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Hydrocortisone; Prednisone; Prednisolone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chronocort® (Experimental): Chronocort® will be provided as 5mg, 10mg and 20mg capsules for oral administration. The starting dose for each subject will be based on the subjects previous glucocorticoid therapy dose and then dose titrated to effect.
  Interventions: Drug: Chronocort®
- standard glucocorticoid therapy (Active Comparator): Subjects in this arm will continue previous oral glucocorticoid therapy titrated to effect.
  Interventions: Drug: standard glucocorticoid therapy

INTERVENTIONS:
Drug: Chronocort® — Chronocort® is a patented oral modified release formulation of hydrocortisone which is intended to mimic, or closely match, the serum levels of endogenous cortisol.
  Other Names: Hydrocortisone
  Arms: Chronocort®
Drug: standard glucocorticoid therapy — Subjects in this arm will continue on their standard hydrocortisone therapy
  Other Names: hydrocortisone; prednisone; prednisolone; dexamethasone
  Arms: standard glucocorticoid therapy

SUMMARY:
This study is a parallel arm, randomised, open-label study, including dose titration and admissions for four overnight stays for 24-hour endocrine profiles. It will compare the efficacy, safety and tolerability of Chronocort® with standard glucocorticoid replacement therapy in the treatment of congenital adrenal hyperplasia (CAH) over a treatment period of 6 months. Dose titration decisions in both treatment groups will be made by a central independent physician, blinded to the treatment arm, using information generated from the 24-hour endocrine profiles. Each treatment arm will be subject to the same titration rules throughout the study, ensuring that opportunities for optimisation and control of androgens are the same in both groups.

DETAILED DESCRIPTION:
At baseline, subjects will be admitted overnight for a 24-hour endocrine profile whilst on their standard therapy. Subjects will attend the study site in the morning and have 17-hydroxyprogesterone (17-OHP) and androstenedione (A4) levels assessed at 15:00, 17:00, 19:00, 21:00, 23:00, 01:00, 03:00, 05:00, 07:00, 09:00, 11:00, 13:00 and 15:00. Safety laboratory tests, a DEXA scan for body composition, and height, weight and waist circumference will be recorded. Subjects will then be randomised to Chronocort® or to continue on their standard care. Randomisation will be stratified by baseline treatment:

1. hydrocortisone only or
2. prednisone or prednisolone, alone or in combination with hydrocortisone
3. dexamethasone only or in combination with any other glucorticoid

The initial dose setting at the start of the Chronocort® treatment will be based on hydrocortisone dose equivalent of baseline therapy in accordance with standard clinical practice. Further dose refinement/titration will be conducted in both treatment groups as necessary after 4 weeks and 12 weeks using a standardised titration algorithm after the subject has been re-admitted for further 24-hour endocrine profiles. Safety endpoints will also be measured at the 07:00 morning sample of each 24-hour profile assessment day. The decision to change doses in both treatment groups will be made by a central independent blinded physician, with the actual change in dose then being made by the local investigator looking after the subject. At 6 months, all the baseline tests will be repeated (including the 24-hour profile). All subjects may then continue on Chronocort®, whatever their randomised treatment, as part of an open-label extension study (to be conducted under a separate protocol). Stress doses of hydrocortisone will be given throughout the study for intercurrent illnesses as medically indicated according to "sick day rules".

ELIGIBILITY:
Inclusion Criteria:

1. Known CAH due to 21-hydroxylase deficiency (classic CAH) diagnosed in childhood with documented (at any time) elevated 17-OHP and/or A4 and currently treated with hydrocortisone, prednisone, prednisolone or dexamethasone (or a combination of the aforementioned glucocorticoids) on a stable glucocorticoid therapy for a minimum of 6 months.
2. Provision of signed written informed consent.
3. Non-pregnant, non-lactating females who are post menopausal, naturally or surgically sterile, or of childbearing potential with a negative urinary pregnancy test and using a medically acceptable method of contraception.
4. Plasma renin activity (PRA) less than 1.5 times the upper limit of normal (ULN) at screening or within 3 months prior to screening, except in subjects who have been diagnosed with hypertension where the renin is not being used to monitor fludrocortisone replacement.
5. Plasma renin activity (PRA) less than 1.5 times the upper limit of normal (ULN) at screening or within 3 months prior to screening, except in subjects who have been diagnosed with hypertension where the renin is not being used to monitor fludrocortisone replacement.

Exclusion Criteria:

1. Co-morbid condition requiring daily administration of a medication (or consumption of any material) that interferes with the metabolism of glucocorticoids.
2. Clinical or biochemical evidence of hepatic or renal disease. Creatinine over twice the ULN or elevated liver function tests (ALT or AST >2 times the ULN).
3. Subjects on regular daily inhaled, topical, nasal or oral steroids for any indication other than CAH.
4. Subjects with any other significant medical or psychiatric conditions that in the opinion of the investigator would preclude participation in the trial.
5. History of malignancy (other than basal cell carcinoma successfully treated >6 months prior to entry into the study).
6. Participation in another clinical trial of an investigational or licensed drug or device within the 3 months prior to inclusion in this study.
7. Subjects with a history of bilateral adrenalectomy.
8. Subjects having previously been exposed to Chronocort®.
9. Subjects unable to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2018-07-28 (Actual); Study Completion 2018-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Merke, MD, Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be decided at a later date

REFERENCES:
- [Derived] Merke DP, Mallappa A, Arlt W, Brac de la Perriere A, Linden Hirschberg A, Juul A, Newell-Price J, Perry CG, Prete A, Rees DA, Reisch N, Stikkelbroeck N, Touraine P, Maltby K, Treasure FP, Porter J, Ross RJ. Modified-Release Hydrocortisone in Congenital Adrenal Hyperplasia. J Clin Endocrinol Metab. 2021 Apr 23;106(5):e2063-e2077. doi: 10.1210/clinem/dgab051. PMID 33527139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 study sites in 7 countries: Denmark 1, France 2, Germany 1,Netherlands 1, Sweden 1, UK 4, and USA 1.
Pre-assignment Details: Following written informed consent and screening tests (Visit 0), eligible participants were called back for the baseline visit. As part of the baseline assessment, participants were admitted overnight for a 24- hour endocrine profile whilst remaining on their standard therapy. Participants were then randomised to Chronocort or standard therapy.
Groups:
- Chronocort®: Chronocort® will be provided as 5mg, 10mg and 20mg capsules for oral administration. The starting dose for each subject will be based on the subject's previous glucocorticoid therapy dose and then dose titrated to effect.
  Chronocort®: Chronocort® is a patented oral modified release formulation of hydrocortisone which is intended to mimic, or closely match, the serum levels of endogenous cortisol.
- Standard Glucocorticoid Therapy: Subjects in this arm will continue their previous oral glucocorticoid therapy, titrated to effect. Standard glucocorticoid therapy may consist of:
  1. Hydrocortisone only
  2. Prednisone or prednisolone, alone or in combination with hydrocortisone
  3. Dexamethasone, alone or in combination with any other glucocorticoid
Period: Overall Study
Arm/Group | Chronocort® | Standard Glucocorticoid Therapy
Started | 61 | 61
Completed | 58 | 59
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronocort® | Standard Glucocorticoid Therapy | Total
Number analyzed (Participants) | 61 | 61 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 59 | 120
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Full Range); unit: years] | 35.2 [19 to 61] | 37.5 [19 to 68] | 36.3 [19 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 36 | 78
  Male | 19 | 25 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 60 | 60 | 120
  Asian | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8
  Europe | 57 | 57 | 114

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 24 Weeks of the Mean of the 24-hour Standard Deviation Score (SDS) Profile for 17-OHP
Description: Change from baseline to 24 weeks of the mean of the 24-hour standard deviation score (SDS) - also referred to as a z-score - profile for 17-OHP (17-Hydroxyprogesterone). The primary efficacy variable was the natural logarithm of the mean of the 24-hour SDS for the natural logarithm of 17-OHP. The mean of the 24-hour SDS profile for each visit was the arithmetic mean of all the SDSs with the first and last (13th) weighted one half relative to the intermediate SDSs. For each of the 13 log-transformed 17-OHP values at each visit, an SDS was calculated by counting the number of SDs that were above or below the mean of the log-transformed range. A negative z-score indicated greater control of 17-OHP when compared to baseline (0).
Time Frame: 24 weeks
Population: The efficacy evaluable analysis set (EES) comprised all participants who were randomised into the study, who received at least one dose of Chronocort or standard GC therapy, and who had an evaluable Week 24 17-OHP 24-hour hormone profile, and who had no major protocol violations. Total sum of participants in the EES = 105.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Chronocort® | Standard Glucocorticoid Therapy
Number analyzed (Participants) | 53 | 52
Z-score | -0.403 (0.8499) | -0.172 (0.7776)
Statistical Analysis 1: Comparison: Chronocort® vs Standard Glucocorticoid Therapy; The primary efficacy variable was the natural logarithm of the mean of the 24-hour SDS profile for the natural logarithm of 17-OHP. The SDS profile was calculated as the SDS of log transformed 17-OHP concentration unsigned. The mean of the 24-hour SDS profile for each visit was the arithmetic mean of all the SDSs, with the first and last (13th) weighted one half relative to the intermediate SDSs; Test type: Superiority; p = 0.5521, ANCOVA; Mean Difference (Final Values) = -0.069, 95% CI 2-sided [-0.299 to 0.161]

2. Secondary Outcome: Change From Baseline to 24 Weeks of the Mean of the 24-hour Standard Deviation Score (SDS) Profile for A4
Description: Change from baseline to 24 weeks of the mean of the 24-hour standard deviation score (SDS) - also referred to as a z-score - profile for A4 (androstenedione). This secondary efficacy variable was calculated as follows: the natural logarithm of the mean of the 24-hour SDS for the natural logarithm of A4. The mean of the 24-hour SDS profile for each visit was the arithmetic mean of all the SDSs with the first and last (13th) weighted one half relative to the intermediate SDSs. For each of the 13 log-transformed A4 values at each visit, an SDS was calculated by counting the number of SDs that were above or below the mean of the log-transformed range. A negative z-score indicated greater control of A4 when compared to baseline (0).
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Chronocort® | Standard Glucocorticoid Therapy
Number analyzed (Participants) | 53 | 52
Z-score | 0.113 (0.9221) | -0.041 (0.7731)
Statistical Analysis 1: Comparison: Chronocort® vs Standard Glucocorticoid Therapy; Change from Baseline to 24 Weeks in A4 Using an ANCOVA Model - The analysis conducted for the primary endpoint variable analysis of 17-OHP was repeated for A4; Test type: Superiority; p = 0.7405, ANCOVA; Mean Difference (Final Values) = 0.047, 95% CI 2-sided [-0.234 to 0.329]

3. Secondary Outcome: 17-OHP and A4 by Individual Baseline Treatment Strata.
Description: 17-OHP and A4 by individual baseline treatment strata presented in the same manner as the primary endpoint (using 24-hour SDS profile at 24 weeks). Change from baseline to 24 weeks of the mean of the 24-hour standard deviation score (SDS) - also referred to as a z-score - profile for 17-OHP and A4. This secondary efficacy variable was calculated as follows: the natural logarithm of the mean of the 24-hour SDS for the natural logarithm of 17-OHP and A4. The mean of the 24-hour SDS profile for each visit was the arithmetic mean of all the SDSs with the first and last (13th) weighted one half relative to the intermediate SDSs. For each of the 13 log-transformed 17-OHP and A4 values at each visit, an SDS was calculated by counting the number of SDs that were above or below the mean of the log-transformed range. A negative z-score indicated greater control of 17-OHP and A4 when compared to baseline (0).
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Pre-Baseline - Hydrocortisone - 17-OHP; Pre-Baseline - Prednisone/Prednisolone - 17-OHP; Pre-Baseline - Dexamethasone - 17-OHP; Pre-Baseline - Chronocort vs. Hydrocortisone - 17-OHP; Pre-Baseline - Chronocort vs. Prednisone/Prednisolone - 17-OHP; Pre-Baseline - Chronocort vs. Dexamethasone - 17-OHP: Secondary efficacy analysis of 17-OHP by pre-treatment strata, change from baseline to 24 weeks in primary efficacy variable, analysis of covariance model (Efficacy evaluable analysis set).
- Pre-Baseline - Hydrocortisone - A4; Pre-Baseline - Prednisone/Prednisolone - A4; Pre-Baseline - Dexamethasone - A4; Pre-Baseline - Chronocort vs. Hydrocortisone - A4; Pre-Baseline - Chronocort vs. Prednisone/Prednisolone - A4; Pre-Baseline - Chronocort vs. Dexamethasone - A4: Secondary efficacy analysis of A4 by pre-treatment strata, change from baseline to 24 weeks in primary efficacy variable, analysis of covariance model (Efficacy evaluable analysis set)
Arm/Group | Pre-Baseline - Hydrocortisone - 17-OHP | Pre-Baseline - Prednisone/Prednisolone - 17-OHP | Pre-Baseline - Dexamethasone - 17-OHP | Pre-Baseline - Chronocort vs. Hydrocortisone - 17-OHP | Pre-Baseline - Chronocort vs. Prednisone/Prednisolone - 17-OHP | Pre-Baseline - Chronocort vs. Dexamethasone - 17-OHP | Pre-Baseline - Hydrocortisone - A4 | Pre-Baseline - Prednisone/Prednisolone - A4 | Pre-Baseline - Dexamethasone - A4 | Pre-Baseline - Chronocort vs. Hydrocortisone - A4 | Pre-Baseline - Chronocort vs. Prednisone/Prednisolone - A4 | Pre-Baseline - Chronocort vs. Dexamethasone - A4
Number analyzed (Participants) | 27 | 21 | 4 | 31 | 18 | 4 | 27 | 21 | 4 | 31 | 18 | 4
Z-score | -0.248 (0.7661) | -0.061 (0.8051) | -0.245 (0.8522) | -0.431 (0.8727) | -0.320 (0.7627) | -0.565 (1.2343) | -0.211 (0.7426) | 0.100 (0.8339) | 0.368 (0.3521) | 0.015 (1.0128) | 0.328 (0.7256) | -0.092 (1.0310)
Statistical Analysis 1: Comparison: Pre-Baseline - Hydrocortisone - 17-OHP vs Pre-Baseline - Chronocort vs. Hydrocortisone - 17-OHP; Test type: Superiority; p = 0.8186, ANCOVA; Mean Difference (Final Values) = -0.037, 95% CI 2-sided [-0.354 to 0.281]
Statistical Analysis 2: Comparison: Pre-Baseline - Prednisone/Prednisolone - 17-OHP vs Pre-Baseline - Chronocort vs. Prednisone/Prednisolone - 17-OHP; Test type: Superiority; p = 0.4655, ANCOVA; Mean Difference (Final Values) = -0.135, 95% CI 2-sided [-0.508 to 0.237]
Statistical Analysis 3: Comparison: Pre-Baseline - Dexamethasone - 17-OHP vs Pre-Baseline - Chronocort vs. Dexamethasone - 17-OHP; Test type: Superiority; p = 0.9081, ANCOVA; Mean Difference (Final Values) = 0.065, 95% CI 2-sided [-1.32 to 1.451]
Statistical Analysis 4: Comparison: Pre-Baseline - Hydrocortisone - A4 vs Pre-Baseline - Chronocort vs. Hydrocortisone - A4; Test type: Superiority; p = 0.6729, ANCOVA; Median Difference (Final Values) = 0.092, 95% CI 2-sided [-0.343 to 0.527]
Statistical Analysis 5: Comparison: Pre-Baseline - Prednisone/Prednisolone - A4 vs Pre-Baseline - Chronocort vs. Prednisone/Prednisolone - A4; Test type: Superiority; p = 0.5322, ANCOVA; Mean Difference (Final Values) = 0.116, 95% CI 2-sided [-0.257 to 0.489]
Statistical Analysis 6: Comparison: Pre-Baseline - Dexamethasone - A4 vs Pre-Baseline - Chronocort vs. Dexamethasone - A4; Test type: Superiority; p = 0.2885, ANCOVA; Mean Difference (Final Values) = -0.568, 95% CI 2-sided [-1.799 to 0.662]

4. Secondary Outcome: Number of Participants With 17-OHP and A4 Levels in the Optimal Range at 9:00 at Week 24 Visit
Description: 17-OHP and A4 levels at 09:00 at the week 24 visit, as a responder analysis (i.e. the number of participants achieving results in the optimal range).
  Optimal range for 17-OHP (male) = 1.2* - 6.7 nmol/L (female) = 1.2* - 8.6 Optimal range for A4 (male) = 1.4 - 5.2 nmol/L (female) = 1.0 - 7.0 nmol/L
  * = There is no lower reference range available for 17-OHP, hence the lower limit of the optimal range was used in the derivation of the average Standard Deviation Score. This enabled calculation of an 'unsigned' SDS score which was used to assess potential over-treatment as well as under-treatment.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Chronocort - 09:00h Response - 17-OHP: Number of participants in the Chronocort arm (from the efficacy evaluable analysis set) achieving 17-OHP levels within the optimal range expected at 09:00h at the week 24 visit.
- Chronocort - 09:00h Response - A4: Number of participants in the Chronocort arm (from the efficacy evaluable analysis set) achieving A4 levels within the optimal range expected at 09:00h at the week 24 visit.
- Standard Glucocorticoid Therapy - 09:00h Response - 17-OHP: Number of participants in the standard glucocorticoid arm (from the efficacy evaluable analysis set) achieving 17-OHP levels within the optimal range expected at 09:00h at the week 24 visit.
- Standard Glucocorticoid Therapy - 09:00h Response - A4: Number of participants in the standard glucocorticoid arm (from the efficacy evaluable analysis set) achieving A4 levels within the optimal range expected at 09:00h at the week 24 visit.
Arm/Group | Chronocort - 09:00h Response - 17-OHP | Chronocort - 09:00h Response - A4 | Standard Glucocorticoid Therapy - 09:00h Response - 17-OHP | Standard Glucocorticoid Therapy - 09:00h Response - A4
Number analyzed (Participants) | 53 | 53 | 52 | 52
Participants | 30 | 25 | 30 | 30
Statistical Analysis 1: Comparison: Chronocort - 09:00h Response - 17-OHP vs Standard Glucocorticoid Therapy - 09:00h Response - 17-OHP; Test type: Superiority; p = 0.9877, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.45 to 2.19]
Statistical Analysis 2: Comparison: Chronocort - 09:00h Response - A4 vs Standard Glucocorticoid Therapy - 09:00h Response - A4; Test type: Superiority; p = 0.8498, Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.43 to 2.02]

5. Secondary Outcome: Changes Relative to Standard Glucocorticoid Therapy in Body Composition (DEXA - Fat Mass and Lean Mass)
Description: Changes relative to Standard glucocorticoid therapy in body composition (DEXA) (fat mass and lean mass) - measured at all sites except Germany.
Time Frame: Baseline and 24 weeks
Population: The efficacy evaluable analysis set (EES) comprised all participants who were randomised into the study, who received at least one dose of Chronocort or standard GC therapy, and who had an evaluable Week 24 17-OHP 24-hour hormone profile, and who had no major protocol violations. German subjects were excluded from this analysis subset.
Measure: Mean (Standard Deviation); unit: kilograms
Groups:
- Chronocort - DEXA - Fat Mass; Standard Glucocorticoid Therapy - DEXA - Fat Mass; Chronocort - DEXA - Lean Mass; Standard Glucocorticoid Therapy - DEXA - Lean Mass: German subjects have been excluded from this analysis group as DEXA scans are not performed at German sites.
Arm/Group | Chronocort - DEXA - Fat Mass | Standard Glucocorticoid Therapy - DEXA - Fat Mass | Chronocort - DEXA - Lean Mass | Standard Glucocorticoid Therapy - DEXA - Lean Mass
Number analyzed (Participants) | 43 | 39 | 43 | 39
kilograms | -0.575 (3.2744) | 0.445 (2.4660) | 0.640 (2.3304) | 0.234 (1.3689)
Statistical Analysis 1: Comparison: Chronocort - DEXA - Fat Mass vs Standard Glucocorticoid Therapy - DEXA - Fat Mass; German subjects have been excluded from this analysis group as DEXA scans are not performed at German sites; Test type: Superiority; p = 0.156, ANCOVA; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-2.294 to 0.374]
Statistical Analysis 2: Comparison: Chronocort - DEXA - Lean Mass vs Standard Glucocorticoid Therapy - DEXA - Lean Mass; German subjects have been excluded from this analysis group as DEXA scans are not performed at German sites; Test type: Superiority; p = 0.3392, ANCOVA; Median Difference (Final Values) = 0.425, 95% CI 2-sided [-0.455 to 1.305]

6. Secondary Outcome: Changes Relative to Standard Glucocorticoid Therapy in Body Composition (DEXA - Bone Mineral Density) - Measured at All Sites Except Germany.
Description: Changes relative to Standard glucocorticoid therapy in body composition (DEXA - bone mineral density only) - measured at all sites except Germany.
Time Frame: Baseline and 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/cm^2
Groups:
- Chronocort - DEXA - Bone Mineral Density; Standard Glucocorticoid Therapy - DEXA - Bone Mineral Density: German subjects have been excluded from this analysis group as DEXA scans are not performed at German sites.
Arm/Group | Chronocort - DEXA - Bone Mineral Density | Standard Glucocorticoid Therapy - DEXA - Bone Mineral Density
Number analyzed (Participants) | 35 | 36
g/cm^2 | -0.001 (0.0250) | -0.008 (0.0399)
Statistical Analysis 1: Comparison: Chronocort - DEXA - Bone Mineral Density vs Standard Glucocorticoid Therapy - DEXA - Bone Mineral Density; Test type: Superiority; p = 0.2614, ANCOVA; Median Difference (Final Values) = 0.009, 95% CI 2-sided [-0.007 to 0.025]

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from the point of enrolment to completion of the study (6 months).
Description: Adverse event information was collected at each visit by the investigator and reported accordingly.
Arm/Group | Chronocort® | Standard Glucocorticoid Therapy
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 7/61 | 5/61
Other Adverse Events (participants affected / at risk) | 59/61 | 48/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronocort® (N=61) | Standard Glucocorticoid Therapy (N=61)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Salpingitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsilitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Adrenocortical Insufficiency (acute) (Endocrine disorders) | 0 (0) | 3 (3)
Adrenal Insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronocort® (N=61) | Standard Glucocorticoid Therapy (N=61)
Acute Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (4)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Tonsilitis (Infections and infestations) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 2 (2)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 12 (16) | 13 (15)
Diarrhoea Infectious (Infections and infestations) | 0 (0) | 1 (1)
Oral Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Otitis Media Acute (Infections and infestations) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (1)
Viral Rash (Infections and infestations) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abnormal Loss of Weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Abnormal Weight Gain (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fluid Retention (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Gluten Sensitivity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperinsulinaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Impaired Fasting Glucose (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Increased Appetite (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Weight Fluctuation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alcohol Intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Affect Lability (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0)
Burnout Syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed Mood (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (6) | 4 (4)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Libido Decreased (Psychiatric disorders) | 1 (1) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 3 (3)
Agitation (Psychiatric disorders) | 0 (0) | 2 (3)
Emotional Distress (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Carpal Tunnel Syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Circardian Rhythm Sleep Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 7 (13) | 4 (5)
Dizziness Postural (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 15 (19) | 15 (22)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral Nerve Lesion (Nervous system disorders) | 1 (1) | 0 (0)
Poor Quality Sleep (Nervous system disorders) | 1 (1) | 0 (0)
Sensory Loss (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (2)
Psychomotor Hyperactivity (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tension Headache (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 3 (3) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Foreign Body Sensation in Eyes (Eye disorders) | 1 (1) | 0 (0)
Lacrimation Increased (Eye disorders) | 1 (1) | 0 (0)
Ear Deformity Acquired (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 3 (3)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (7) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric Discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (9) | 4 (5)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (4)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum Intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces Soft (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cold Sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hair Growth Abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chloasma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Menstruation Irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 4 (6) | 3 (3)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Fat Tissue Increased (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 9 (13) | 10 (20)
Inflammation (General disorders) | 1 (1) | 0 (0)
Influenza-like Illness (General disorders) | 2 (3) | 4 (4)
Malaise (General disorders) | 5 (5) | 2 (2)
Pyrexia (General disorders) | 9 (9) | 4 (4)
Therapeutic Response Unexpected (General disorders) | 10 (15) | 1 (1) — AE of unexpected therapeutic benefit
Thirst (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (3)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1)
Sensation of Foreign Body (General disorders) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Blood Sodium Decreased (Investigations) | 1 (1) | 0 (0)
Body Temperature Increased (Investigations) | 2 (2) | 0 (0)
Osteocalcin Decreased (Investigations) | 1 (1) | 0 (0)
Renin Increased (Investigations) | 3 (3) | 7 (7)
Urine Output Decreased (Investigations) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 1 (1)
Blood Glucose Increased (Investigations) | 0 (0) | 1 (1)
C-Telopeptide Increased (Investigations) | 0 (0) | 1 (1)
Haematocrit Decreased (Investigations) | 0 (0) | 1 (1)
Haemoglobin Decreased (Investigations) | 0 (0) | 1 (1)
Liver Function Test Abnormal (Investigations) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 0 (0) | 1 (1)
White Blood Cell Count Increased (Investigations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Auricular Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ear Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mineralocorticoid Deficiency (Endocrine disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 3 (3)
Salpingitis (Infections and infestations) | 1 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
A limitation of the pre-defined primary endpoint was that it included an unsigned SDS score over a 24-hour period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Specified in the contractual agreements between the Sponsor and investigators: "Neither the CRO, nor the Heath Board, nor the Investigator shall register the Clinical Trial, or the results, on any publicly accessible clinical trial registry."

DOCUMENTS (2):
  • Study Protocol (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT02716818/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT02716818/SAP_001.pdf